CLINICAL TRIAL: NCT05608577
Title: RE-BLEED: A Digital Platform for Identifying Bleeding Patients - a Feasibility Study
Acronym: RE-BLEED
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: University of Leicester (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PID15451
Record Dates: First submitted 2022-10-21; First posted 2022-11-08 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Hemorrhage; Trauma; Gastro Intestinal Bleeding
MeSH Terms: conditions — Hemorrhage; Wounds and Injuries; Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Ethylenediamine tetraacetic acid (and citrate blood samples taken as part of routine clinical care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: Up to 1,750,000 patient admissions (up to 10 years of admissions) from one National Health Service Trust (Hospital group)
- Prospective Hospital Cohort: Up to 87, 500 will be screened by the digital platform to identify those who may have bled during the recruitment period, of which at least 40 will be approached for their consent to retain their blood samples (collected as part of routine care).

SUMMARY:
The RE-BLEED feasibility study aims to develop and test a real-time digital platform, whereby bleeding patients in-hospital can be identified and approached for their consent to participate in future research studies.

DETAILED DESCRIPTION:
Bleeding affects up to 40% of all trauma patients, up to 30% of all surgery patients and is one of the commonest causes of death for women giving birth. The presentation and features of bleeding are different between patients - in some cases bleeding is very obvious to recognise, but in other cases bleeding is more "hidden", for example in the stomach. Bleeding must be stopped promptly to prevent severe illness or death.

Many studies have shown differences in how patients who bleed are treated. There is also variation in how individual patients respond to the same treatment, with some patients doing better than others. Understanding how variation in practice and patient characteristics affect outcomes will help researchers and clinicians design and test improvements in care.

Patients in hospital have regular tests that measure levels of the different types of cells in their blood and its ability to clot. For example, a drop in red blood cells can indicate that patients have suffered bleeding. More advanced blood tests are available that can provide more detailed information on why patients are bleeding and what treatments might be most effective.

This study aims to develop a real-time, hospital-wide digital system to identify patients in hospital who have suffered from bleeding and test whether this system could be used in the future to potentially identify patients to recruit into trials of new treatments or blood tests.

To do this, the investigators will:

* Assemble a panel of experts to identify criteria (for example, specific blood test results and drug prescriptions) that could indicate a patient has suffered from bleeding
* Use historical electronic patient records to test how well these criteria identify patients who have received treatments for bleeding (blood transfusion)
* Develop and refine a web-based digital system where the most useful criteria can be applied in "real-time" to identify bleeding patients
* Test how well the digital platform identifies bleeding patients
* Test whether a significant number of patients identified by the digital platform are willing to allow their routine blood samples tested for blood clotting and endothelial factors.

ELIGIBILITY:
Inclusion Criteria:

Retrospective cohort:

* Adults aged between 16 and 110
* Admitted to hospital (Oxford University Hospitals NHS Foundation Trust) or attended the emergency department between 1/3/2011 to 31/8/2023

Prospective cohort:

* Adults aged between 16 and 110
* Admitted to hospital (Oxford University Hospitals NHS Foundation Trust) or attended the emergency department between 1/10/2021 to 31/8/2023

Exclusion Criteria:

Both retrospective and prospective cohorts:

* Patients who inform us directly that they do not wish their records used in this research study
* Patients who have completed the NHS Opt-out.

Ages: 16 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult patients admitted to Oxford University Hospitals NHS Foundation Trust
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Within 3 months from start of recruitment
  Number of patients identified who consent for their blood samples to be retained and analysed as a percentage of those correctly identified as having suffered bleeding by the REBLEED system.
  An acceptable recruitment rate is defined as at least 20%, from a total of at least 200 patients correctly identified as having suffered bleeding by the REBLEED system.
  Patients correctly identified as having suffered bleeding by the REBLEED system is defined as: Flagged by REBLEED system as potentially having suffered bleeding AND confirmed as having suffered bleeding by research nurse review of electronic medical records

CONTACTS AND LOCATIONS:
Overall Officials: Peter Watkinson, MD, Principal Investigator — University of Oxford
Locations (1):
- Oxford University Hospitals NHS Foundation Trust (John Radcliffe Hospital), Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made publicly available due to privacy and legal implications.

DOCUMENTS (1):
  • Study Protocol (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT05608577/Prot_000.pdf